CLINICAL TRIAL: NCT02929355
Title: Progression of Carotid Atherosclerosis and Vascular Events in People With Diabetes: A Prospective Cohort Study
Brief Title: Carotid Atherosclerosis and Vascular Events in People With Diabetes
Acronym: PROCAVE-D
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0596
Record Dates: First submitted 2016-09-23; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-09

CONDITIONS: Carotid Atherosclerosis
Keywords: Carotid atherosclerosis; duplex ultrasonography; diabetes; vascular events
MeSH Terms: conditions — Carotid Artery Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diabetic patients with carotid assessment: Patients with diabetes and a carotid assessment by duplex ultrasonography in 2012 in a monocentric diabetic unit
  Interventions: Other: carotid assesment by duplex ultrasonography

INTERVENTIONS:
Other: carotid assesment by duplex ultrasonography

SUMMARY:
Diabetes is a risk factor for carotid atherosclerotic whose progression is associated with an increased risk of vascular events. Investigators assessed prospectively by arterial duplex ultrasonography the progression of carotid atherosclerosis in a cohort of people with diabetes to assess the importance of progression and to analyze the impact of this progression on vascular events. The main hypothesis is that people with carotid atherosclerosis progression are at higher risk of vascular events than those without any progression.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 ans
* Diabetes
* Carotid duplex ultrasonography in 2012

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes and a carotid assessment by duplex ultrasonography in 2012 in a monocentric diabetic unit
Sampling Method: Non-Probability Sample
Enrollment: 731 (Actual)
Dates: Start 2012-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Rate of vascular events between day one and the last day of follow-up reviewed by patient examination | Day of the last assessment of carotid atherosclerosis by duplex ultrasonography (between 01/2014 and 09/2016)
  Vascular events include ischemic myocardial events, ischemic cerebrovascular events, lower limb ischemia, arterial revascularization procedure

SECONDARY OUTCOMES:
Rate of carotid atherosclerosis progression measured by duplex ultrasonography in percentage of stenosis | Day of the last assessment of carotid atherosclerosis by duplex ultrasonography between 01/2014 and 09/2016.
  At each visit, carotid arteries were examined by duplex ultrasonography. The most severe lesion for each patient was selected. Results were classified in three Strandness categories: normal (no atherosclerotic lesions), stenosis < 50% (systolic ratio Internal Carotid Artery (ICA)/Common Carotid Artery (CCA) < 2) and stenosis ≥ 50% (systolic ratio ICA/CCA ≥ 2). A progression was the move to a higher category.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Endocrinologie, Diabète et Maladie de la Nutrition, GH Sud, Hospices Civils de Lyon, Pierre-Bénite, France

REFERENCES:
- [Derived] Vouillarmet J, Marsot C, Maucort-Boulch D, Riche B, Helfre M, Grange C. Vascular Events and Carotid Atherosclerosis: A 5-Year Prospective Cohort Study in Patients with Type 2 Diabetes and a Contemporary Cardiovascular Prevention Treatment. J Diabetes Res. 2019 Dec 22;2019:9059761. doi: 10.1155/2019/9059761. eCollection 2019. PMID 31934592